CLINICAL TRIAL: NCT00583609
Title: A Pilot Study of a New PEG3350 Dose Formulation For Use in Constipated Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: John McGowan, Clinical Operations Manager, Braintree Laboratories, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851-PP-03
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PEG3350
  Interventions: Drug: PEG3350

INTERVENTIONS:
Drug: PEG3350 — PEG3350

SUMMARY:
To evaluate the patient acceptance of a new PEG3350 dose formulation in children currently treated with PEG3350 powder for treatment of constipation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female constipated outpatients between the ages of 4 and 16
* Currently taking a dose of PEG 3350 powder up to a maximum of 17g per day that has been consistent for at least 4 weeks, or if less than 4 weeks, the investigator testifies that the patient is stable
* Current treatment is considered successful - defined as greater than 2 bowel movements per week with no accidents
* Are otherwise in good health, as judged by a physical examination
* If female and of childbearing potential, patient must be using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so for the duration of the study
* In the investigator's judgment, patient or guardian is mentally competent to sign an instrument of informed consent

Exclusion Criteria:

* Patients who are impacted at baseline exam
* Patients with known or suspected perforation or obstruction
* Patients with a history of gastric retention, inflammatory bowel disease, bowel resection, or colostomy
* Patients with a known history of organic cause for their constipation
* Patients currently using medications known to cause constipation (these include opiates, antidepressants, SSRI's, antimotility agents and anticholinergics)
* Patients who are breastfeeding, pregnant, or intend to become pregnant during the study
* Female patients of childbearing potential who refuse a pregnancy test
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedure
* Patients with known allergy to PEG or PEG containing medications
* Patients who, within the past 30 days have participated in an investigational clinical study

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Efficacy will be measured by analysis of patient self reported bowel movement (BM) data | 2 weeks

SECONDARY OUTCOMES:
Adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (2):
- United States (2):
  - Little Rock, Arkansas
  - Morristown, New Jersey